CLINICAL TRIAL: NCT06189950
Title: a Prospective, Multi-center, Open-label, Non-inferiority, Randomized, Controlled Registration Trial of the Intracranial Stent for the Treatment of Intracranial Aneurysms: Rebridge
Brief Title: Registration Trial of the Intracranial Visualized Stent for the Wide-necked Intracranial Aneurysms:REBRIDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mermaid-2023-01-CIP-00
Record Dates: First submitted 2023-12-14; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Brain Diseases; Aneurysm; Intracranial Aneurysm
MeSH Terms: conditions — Brain Diseases; Aneurysm; Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Microport NeuroTech Intracranial Visualized Stent
  Interventions: Device: Intracranial stent for wide-necked aneurysms
- Control group (Active Comparator): LVIS™ and LVIS™ Jr
  Interventions: Device: Intracranial stent for wide-necked aneurysms

INTERVENTIONS:
Device: Intracranial stent for wide-necked aneurysms — Intracranial stent for wide-necked aneurysms

SUMMARY:
This trial was designed as a prospective, multicentre, open, non-inferiority, randomised controlled clinical trial, with the control devices being MicroVention's LVIS Intraluminal Support Device and LVIS Jr. Intraluminal Support Device. Approximately 200 subjects with intracranial aneurysms would be enrolled for stent-assisted coiling embolisation according to the inclusion and exclusion criteria specified in this trial protocol. Subjects were evaluated by mRS preoperatively, at the time of device implantation, at the time of discharge from the hospital, at 1 month (±7 days) postoperatively, at 6 months (±30 days) postoperatively, and at 12 months (±60 days) postoperatively; subjects would underwent DSA imaging at surgery and at 6 months (±30 days) postoperatively, and MRA or DSA imaging at 12 months (±60 days) postoperatively. Unplanned follow-up of the subjects would performed when necessary, and data would be recorded to evaluate the safety and efficacy of intracranial artery stent for stent-assisted coiling embolisation for the treatment of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent form(ICF), the applicant shall be male or non-pregnant female, aged 18 to 80 years； Target aneurysms was diagnosed as intracranial widenecked saccular aneurysms by DSA/CTA/MRA； The target aneurysm should be suitable for stentassisted coiling surgery and could be treated through one operation； Subject or its legal representative should be able to understand the purpose of this study, also agree to comply with protocol and sign the informed consent form voluntarily.

Exclusion Criteria:

* Aneurysms unsuitable for stent-assisted coiling (i.e. aneurysm necks ≤ 4 mm and or body-to-neck ratio ≥ 2)； The distal diameter of the aneurysm-carrying artery is outside the range of application of the investigational device; mRS score ≥3; Subjects with recurrent aneurysms treated by stent-assisted coiling; Multiple aneurysms and all aneurysms requiring intervention; Subjects with ruptured aneurysms <30 days ; Significant stenosis (≥50%) or occlusion of parent artery; Subjects unsuitable for anaesthesia or endovascular surgical treatment, e.g. major diseases of the heart, lungs, liver, spleen and kidneys, brain tumours, severe active infections, disseminated intravascular coagulation, and a history of severe mental illness; Subjects undergoing major surgical procedures (e.g. tumour resection, surgery of vital organs, etc.) within 30 days prior to signing the informed consent form, or scheduled to undergo such procedures within 60 days after signing the informed consent form; Subjects with morphologies or pathologies that may interfere with device use, including, but not limited to: carotid artery coarctation, vasculitis, aortic coarctation, limited vascular access (e.g., severe intracranial vascular tortuosity, severe intracranial vasospasm unresponsive to medication, other anatomical or clinical pathologies that would prevent access to the device); Contraindications to stenting, including but not limited to: contraindication to DSA, allergy or intolerance to contrast media, allergy or intolerance to antiplatelet and anticoagulant medications required for treatment, allergy to nickel-titanium and platinum-tungsten and platinum-iridium alloys; Pregnant or breastfeeding women; Life expectancy less than 12 months; Subject participation in other drug or device studies that do not meet endpoints

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Rate of aneurysms with adequate occlusion | 6 months
  The Raymond-Roy intracranial aneurysm occlusion classification was used to assess the rate of aneurysm occlusion postoperatively or at the time of primary endpoint assessment (12 months). Occlusion rates were reported as Class I: complete occlusion; Class II: residual neck; Class III: residual aneurysm.
  Adequate occlusion rate includes Class I and Class II

SECONDARY OUTCOMES:
Rate of stent technical success | immediately after the procedure
  Technical successwas defined as the stent was successfully released at the appropriate position, and covered the aneurysm's neck completely while the parent artery remained unobstructed postoperatively.
Rate of aneurysms with complete occlusion | 6 months
  The Raymond-Roy intracranial aneurysm occlusion classification was used to assess the rate of aneurysm occlusion postoperatively or at the time of primary endpoint assessment (12 months). Occlusion rates were reported as Class I: complete occlusion; Class II: residual neck; Class III: residual aneurysm.
  Complete occlusion rate includes Class I
Rate of in-stent stenosis (≥50%) | 6 months
Rate of aneurysms with adequate occlusion | 1 year
Rate of aneurysms with complete occlusion | 1 year
Rate of aneurysms with retreatment | 1 year
  Percentage of subjects who had aneurysm recurrence and underwent a secondary suergry during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: sheng guan, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No